CLINICAL TRIAL: NCT05293743
Title: Development and Evaluation of Novel Dynamic Bar for Foot Abduction Brace for Clubfoot Treatment
Brief Title: Novel Dynamic Foot Abduction Bar for Treatment of Clubfoot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Maryse Bouchard, Assistant Professor, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Device Feasibility
Other Study IDs: 1000078967
Record Dates: First submitted 2021-10-31; First posted 2022-03-24 (Actual); Results first posted 2024-11-25 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Clubfoot
MeSH Terms: conditions — Clubfoot

STUDY DESIGN:
Intervention Model Description: Experimental arm with new device, control arm with standard device.
Who Masked: Outcomes Assessor
Masking Description: The clinician assessing foot shape for recurrence will be blinded to the brace type. Clinicians involved in fitting the brace will not be.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Bar (Active Comparator): This group will continue using the Standard Bar as part of their brace, per their current treatment.
  Interventions: Device: Foot abduction bracing for clubfoot with Standard Bar
- Dynamic Bar (Experimental): This group will use the Dynamic Bar for 30 days instead of their Standard Bar.
  Interventions: Device: Foot abduction bracing for clubfoot with novel Dynamic Bar

INTERVENTIONS:
Device: Foot abduction bracing for clubfoot with novel Dynamic Bar — After Ponseti treatment of serial casting and tenotomy for clubfoot, patients are braced full time x 3 months then night time until age 5. This study compares standard bars in a foot abduction brace to our novel Dynamic Bar. This group uses the Dynamic Bar.
  Arms: Dynamic Bar
Device: Foot abduction bracing for clubfoot with Standard Bar — After Ponseti treatment of serial casting and tenotomy for clubfoot, patients are braced full time x 3 months then night time until age 5. This study compares standard bars in a foot abduction brace to our novel Dynamic Bar. This group uses the Standard Bar.
  Arms: Standard Bar

SUMMARY:
The goal of this clinical trial is to evaluate a new Dynamic Bar for foot abduction bracing for clubfoot treatment. The main questions that this study aims to answer are:

* How easy is it to recruit and retain participants for a randomized-controlled effectiveness trial of a novel foot abduction bar?
* How does parental perception of child comfort in the Dynamic Bar compare to parental perception of child comfort in standard bars?
* How does patient tolerance of the Dynamic Bar compare patient tolerance of standard bars?
* How effective is the Dynamic Bar at preventing clubfoot recurrence during the bracing phase when the brace is worn as prescribed for a 30-day trial period?

Each participant will be randomized into one of two arms: the experimental arm or the control arm. For the first 30 days, the experimental arm will wear the new Dynamic Bar with standard boots and the control arm will continue wearing their standard bar. After this 30-day period, the experimental arm will return to wearing their standard bar.

DETAILED DESCRIPTION:
This is an assessor-blinded randomized feasibility trial assessing the feasibility of conducting a large-scale clinical trial to evaluate the effectiveness of a new dynamic bar for foot abduction bracing for clubfoot treatment. Feasibility will be determined by the ability to recruit patients within the goal study period and to retain participants. Eligible patients must have a well-corrected idiopathic clubfoot (Pirani Score ≤ 0.5) and be in the minimum 12 hours per day bracing stage of the Ponseti clubfoot treatment protocol. The overall study period will be 90 days in length. For the first 30 days, the experimental cohort will wear the new Dynamic Bar (DB) with standard ankle-foot orthoses (boots) and the control cohort will continue wearing their Standard Bar (SB). After this 30-day period, the experimental cohort will return to wearing their SB.

All patients will be evaluated on Day 0, Day 7, Day 30, and Day 90 of the study period to monitor for recurrence of the clubfoot deformity, complications of brace wearing, to submit brace wear logs, and to complete parent-reported questionnaires regarding their perceptions of the Foot Abduction Brace (FAB) and their child's comfort. A minimum of 10 patients per arm will be recruited. A temperature sensor will be added in each participant's boots during the 90-day study period to objectively measure time of brace wear. It is hypothesized that when patients are wearing the DB, they will experience higher brace tolerance defined as increased wear time of the brace as measured by the temperature sensors, and higher comfort levels as reported by parents, without an increase in clubfoot deformity recurrence compared to the SB.

Most patient information that will be reviewed in this study is data being collected and stored per the REB-approved Clubfoot Research Registry protocol (REB #1000053919). All patients enrolled in study this will also be enrolled in Clubfoot Research Registry, if not already enrolled.

The novel DB is designed by the research team and allows independent movement of the knees and hips while maintaining a corrective position of the foot.

ELIGIBILITY:
Inclusion Criteria:

1. Ability of parent/care giver to complete brace wear log/surveys in English
2. Diagnosis of idiopathic clubfoot (unilateral or bilateral).
3. Current use of a SB with their Foot Abduction Brace.
4. In the minimum 12-hour per day bracing stage of the Ponseti treatment
5. Aged 1 to 3 years (as the DB prototype was designed based on the average size and strength of a child within that age group).
6. Well-corrected clubfoot/clubfeet (Pirani score ≤ 0.5)
7. Enrollment in the SickKids Clubfoot Research Registry.

Exclusion Criteria:

1. Recurrent clubfoot deformity at time of recruitment and/or Day 0 in study period: Pirani score above 0.5; Presence of cavus, adduction, or hindfoot varus; Less than 10 degrees of passive ankle dorsiflexion.
2. Current complaint of significant brace intolerance.
3. Any condition or diagnosis, that could in the opinion of the Principal Investigator or delegate interfere with the participant's ability to comply with study instructions, might confound the interpretation of the study results, or put the participant at risk, i.e., skin conditions such as eczema, neurologic conditions or any non-idiopathic clubfoot, any acute or chronic illness perceived to be causing the child discomfort such as a cold or flu or other concurrent painful procedure.
4. The patient does not adequately fit the available prototype, e.g., shoulder width distance is too narrow or wide for prototype bar width. However, these patients will be recorded in the study enrollment log to identify the size of this subset. The age and fit issues of these patients will also be recorded to allow future adaptations of the new DB to accommodate this subset.
5. The patient is using an older boot model, in which a temperature sensor cannot be inserted, and the patient does not adequately fit the available boots, in which the temperature sensors have already been installed.

Ages: 1 Year to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2022-08-17 (Actual); Primary Completion 2023-05-24 (Actual); Study Completion 2023-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maryse Bouchard, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
We do not plan on sharing this data with other researchers.

REFERENCES:
- [Background] Anand A, Sala DA. Clubfoot: etiology and treatment. Indian J Orthop. 2008 Jan;42(1):22-8. doi: 10.4103/0019-5413.38576. PMID 19823650
- [Background] Alves C. Bracing in clubfoot: do we know enough? J Child Orthop. 2019 Jun 1;13(3):258-264. doi: 10.1302/1863-2548.13.190069. PMID 31312265
- [Background] Hospital for Special Surgery [Internet]. New York: HSS. Method for Correcting Clubfoot: Overview for Parent; 2019 Sept 12 [cited 2021 Jan 11] Available from: https://www.hss.edu/conditions_thse-ponseti-method-for-clubfoot-correction.asp.
- [Background] Garg S, Porter K. Improved bracing compliance in children with clubfeet using a dynamic orthosis. J Child Orthop. 2009 Aug;3(4):271-6. doi: 10.1007/s11832-009-0182-9. Epub 2009 Jun 3. PMID 19495824
- [Background] SickKids Internal Document. CLUBFOOT FAO BAR OPTIONS June 2017 edited. 2017 June.
- [Background] Azarpira MR, Emami MJ, Vosoughi AR, Rahbari K. Factors associated with recurrence of clubfoot treated by the Ponseti method. World J Clin Cases. 2016 Oct 16;4(10):318-322. doi: 10.12998/wjcc.v4.i10.318. PMID 27803913
- [Background] Zhao D, Liu J, Zhao L, Wu Z. Relapse of clubfoot after treatment with the Ponseti method and the function of the foot abduction orthosis. Clin Orthop Surg. 2014 Sep;6(3):245-52. doi: 10.4055/cios.2014.6.3.245. Epub 2014 Aug 5. PMID 25177447
- [Background] American Academy of Orthopaedic Surgeons [Internet]. Illinois: AAOS. Study Finds Ponseti Method Remains an Effective Treatment for Clubfoot, Bracing Is Paramount; 2021 Jan 18 [cited 2021 May 25] Available from: https://www.aaos.org/aaosnow/2020/aaos-now-special-edition/research/662_pediatrics.
- [Background] Gelfer Y, Wientroub S, Hughes K, Fontalis A, Eastwood DM. Congenital talipes equinovarus: a systematic review of relapse as a primary outcome of the Ponseti method. Bone Joint J. 2019 Jun;101-B(6):639-645. doi: 10.1302/0301-620X.101B6.BJJ-2018-1421.R1. PMID 31154846
- [Background] Morgenstein A, Davis R, Talwalkar V, Iwinski H Jr, Walker J, Milbrandt TA. A randomized clinical trial comparing reported and measured wear rates in clubfoot bracing using a novel pressure sensor. J Pediatr Orthop. 2015 Mar;35(2):185-91. doi: 10.1097/BPO.0000000000000205. PMID 24787312
- [Background] Aroojis A, Pandey T, Dusa A, Krishnan AG, Ghyar R, Ravi B. Development of a functional prototype of a SMART (Sensor-integrated for Monitoring And Remote Tracking) foot abduction brace for clubfoot treatment: a pre-clinical evaluation. Int Orthop. 2021 Sep;45(9):2401-2410. doi: 10.1007/s00264-021-05042-0. Epub 2021 Apr 22. PMID 33885922
- [Background] Sangiorgio SN, Ho NC, Morgan RD, Ebramzadeh E, Zionts LE. The Objective Measurement of Brace-Use Adherence in the Treatment of Idiopathic Clubfoot. J Bone Joint Surg Am. 2016 Oct 5;98(19):1598-1605. doi: 10.2106/JBJS.16.00170. PMID 27707845
- [Background] Masrouha KZ, Moses MJ, Sala DA, Litrenta J, Lehman WB, Chu A. The Validity of Patient-reported Outcome Measurement Information System (PROMIS) Parent Proxy Instruments to Assess Function in Children With Talipes Equinovarus. J Pediatr Orthop. 2019 Nov/Dec;39(10):e787-e790. doi: 10.1097/BPO.0000000000001368. PMID 30913133
- [Background] Varni JW, Limbers CA, Burwinkle TM. How young can children reliably and validly self-report their health-related quality of life?: an analysis of 8,591 children across age subgroups with the PedsQL 4.0 Generic Core Scales. Health Qual Life Outcomes. 2007 Jan 3;5:1. doi: 10.1186/1477-7525-5-1. PMID 17201920
- [Background] Mitchell JR, inventor. Quick clip for a club foot device. United States patent US 20160113803A1. 2002 Jun 9.
- [Background] C-Pro Direct [Internet]. Ponseti AFO Standard Sandals with Bar; [cited 2021 May 25] Available from: https://c-prodirect.com/ponseti-afo-standard-sandals-with-bar.
- [Background] MD Orthopaedics [Internet]. Massachusetts: MD Orthopaedics. Ponseti® Bar; [cited 2021 May 25] Available from: https://mdorthopaedics.easyordershop.com/link/en/bars/ponseti/a/.
- [Background] iButtonLink Technology [Internet]. DS1922L-F5# Thermochron iButton 8K -40 to 85°C; [cited 2021 July 1] Available from: https://www.ibuttonlink.com/products/ds1922l.
- [Background] Dobbs MB, Frick SL, Mosca VS, Raney E, VanBosse HJ, Lerman JA, Talwalkar VR, Steger-May K, Gurnett CA. Design and descriptive data of the randomized Clubfoot Foot Abduction Brace Length of Treatment Study (FAB24). J Pediatr Orthop B. 2017 Mar;26(2):101-107. doi: 10.1097/BPB.0000000000000387. PMID 27632641
- [Background] Tamarack Habilitation Technologies, Inc. [Internet] ShearBan® Self-Adhesive, Low-Friction Sheets for Foot Blister and Ulcer Care; [cited 2021 August 2] Available from: https://tamarackhti.com/resources/shearban
- [Background] Youtube [Internet]. Installing I-Button in Ponseti AFO; [cited 2021 July 1] Available from: https://www.youtube.com/watch?v=YACSbFn-lOA.
- [Background] Sadler B, Gurnett CA, Dobbs MB. The genetics of isolated and syndromic clubfoot. J Child Orthop. 2019 Jun 1;13(3):238-244. doi: 10.1302/1863-2548.13.190063. PMID 31312262
- [Background] D-Bar Enterprises [Internet]. Missouri: D-Bar Enterprises. Product Guide and Catalog ® Bar; 2015 [cited 2021 May 27] Available from: https://www.dobbsbrace.com/products.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at the Clubfoot Clinic in the Hospital for Sick Children between August 2022 and March 2023. The first participant was enrolled on August 17, 2022, and the last participant was enrolled on February 15, 2023.
Pre-assignment Details: Out of the 17 participants who consented to participate, 5 withdrew before beginning their participation in the study. The remaining 12 participants were randomized to treatment, however 1 control participant withdrew after their first study visit.
Groups:
- Control Arm: This group continued using the Standard Bar as part of their brace, per their current treatment.
- Experimental Arm: This group used the Dynamic Bar for 30 days instead of their Standard Bar.
Period: Overall Study
Arm/Group | Control Arm | Experimental Arm
Started | 5 | 7
Completed | 4 | 7
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Arm | Experimental Arm | Total
Number analyzed (Participants) | 4 | 7 | 11
Age, Continuous [Mean (Full Range); unit: months] — Eligible patients had to be over the age of 1 and under the age of 4 at the time of consent (>12 months and <48 months).
  months | 24.9 [16 to 36] | 27.6 [15.5 to 46.5] | 26.6 [15.5 to 46.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 4 | 5 | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Diagnosis [Count of Participants; unit: Participants]
  Unilateral idiopathic clubfoot | 3 | 5 | 8
  Bilateral idiopathic clubfoot | 1 | 2 | 3
Height [Mean (Full Range); unit: cm] | 87.7 [81.5 to 95] | 89.9 [80.5 to 105] | 89.1 [80.5 to 105]
Weight [Mean (Full Range); unit: kg] | 13.5 [11 to 15.8] | 13.9 [10.8 to 19.9] | 13.8 [10.8 to 19.9]

OUTCOME MEASURES:

1. Primary Outcome: Recruitment of Patients for a Prospective Trial Comparing Clubfoot Brace Types
Description: The study's recruitment rate was calculated to evaluate the ease of recruiting participants for a randomized-controlled effectiveness trial of a novel foot abduction bar. A recruitment rate less than 50% is considered a poor indicator for ease of recruitment and protocols for a future study should be revisited to improve recruitment strategies.
Time Frame: Recruitment period lasted approximately 8 months.
Population: 79 patients were deemed eligible to participate and approached for consent during the recruitment period.
Measure: Count of Participants; unit: Participants
Groups:
- Expected Number of Patients Recruited: Number of eligible patients who were expected to consent to participate.
- Actual Number of Patients Recruited: Number of eligible patients who did consent to participate.
Arm/Group | Expected Number of Patients Recruited | Actual Number of Patients Recruited
Number analyzed (Participants) | 79 | 79
Participants | 59 | 17

2. Primary Outcome: Retention of Patients for a Prospective Trial Comparing Clubfoot Brace Types
Description: The dropout rate was calculated to evaluate the ease of retaining participants for a randomized-controlled effectiveness trial of a novel FAB bar. A dropout rate greater than 20% is considered a poor indicator for ease of participant retention.
Time Frame: Study period lasted approximately 90 days.
Population: 17 patients initially consented to participate in the study.
Measure: Count of Participants; unit: Participants
Groups:
- Expected Number of Dropouts: Number of participants who were expected to withdraw from the study after consenting to participate.
- Actual Number of Dropouts: Number of participants who did withdraw from the study after consenting to participate.
Arm/Group | Expected Number of Dropouts | Actual Number of Dropouts
Number analyzed (Participants) | 17 | 17
Participants | 0 | 6

3. Primary Outcome: Parent Satisfaction in a Prospective Trial Comparing Clubfoot Brace Types
Description: On the first day of the study, parents were asked in a questionnaire if they had any concerns about participating in the study. On the last day of the study, parents were asked if they would be interested in participating in a future study of the Dynamic Bar.
  These questions were asked to evaluate the ease of achieving parent satisfaction during a randomized-controlled effectiveness trial of a novel FAB bar.
Time Frame: Study period lasted approximately 90 days.
Population: 4 patients completed participation in the control arm, and 7 patients completed participation in the experimental arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Control Arm | Experimental Arm
Number analyzed (Participants) | 4 | 7
Participants
  First day: Parents asked if they had concerns about participating in the study.: Strongly Disagree | 1 | 3
  First day: Parents asked if they had concerns about participating in the study.: Disagree | 3 | 4
  First day: Parents asked if they had concerns about participating in the study.: Unsure | 0 | 0
  First day: Parents asked if they had concerns about participating in the study.: Agree | 0 | 0
  First day: Parents asked if they had concerns about participating in the study.: Strongly Agree | 0 | 0
  Last day: Parents asked if they would be interested in participating in a future study.: Strongly Disagree | 0 | 0
  Last day: Parents asked if they would be interested in participating in a future study.: Disagree | 0 | 0
  Last day: Parents asked if they would be interested in participating in a future study.: Unsure | 0 | 1
  Last day: Parents asked if they would be interested in participating in a future study.: Agree | 2 | 1
  Last day: Parents asked if they would be interested in participating in a future study.: Strongly Agree | 2 | 5

4. Secondary Outcome: Parental Perception of Child Comfort - How the Dynamic Bar Compares to the Standard Bar
Description: On the last day of the study, parents in the experimental arm were asked in a questionnaire how they thought the Dynamic Bar compared to their original bar, regarding their child's comfort. This was asked to compare parental perception of child comfort in the Dynamic Bar to the Standard Bar.
Time Frame: Study period lasted approximately 90 days.
Population: 7 participants were randomized to the experimental arm to try out the Dynamic Bar.
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Arm
Number analyzed (Participants) | 7
Participants
  Much less comfortable | 0
  Less comfortable | 0
  Equally comfortable | 0
  More comfortable | 4
  Much more comfortable | 3

5. Secondary Outcome: Parental Perception of Child Comfort - Preferred Bar
Description: Parents in the experimental arm were asked to indicate their preferred bar for clubfoot bracing at two different points during the study. This was asked to compare parental perception of child comfort in the Dynamic Bar to the Standard Bar.
Time Frame: Parents were asked to indicate their preferred bar for clubfoot bracing at the end of the study's intervention period (after approximately 30 days) and on the last day of the study (after approximately 90 days).
Population: 7 participants were randomized to the experimental arm to try out the Dynamic Bar.
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Arm
Number analyzed (Participants) | 7
Participants
  Parent asked to indicate their preferred bar at the end of the study's intervention period.: Standard Bar | 0
  Parent asked to indicate their preferred bar at the end of the study's intervention period.: Unsure | 2
  Parent asked to indicate their preferred bar at the end of the study's intervention period.: Dynamic Bar | 5
  Parent asked to indicate their preferred bar at the end of the study's intervention period.: Other | 0
  Parent asked to indicate their preferred bar on the last day of the study.: Standard Bar | 0
  Parent asked to indicate their preferred bar on the last day of the study.: Unsure | 1
  Parent asked to indicate their preferred bar on the last day of the study.: Dynamic Bar | 6
  Parent asked to indicate their preferred bar on the last day of the study.: Other | 0

6. Secondary Outcome: Parental Perception of Child Comfort - If Child Had a Hard Time Returning to the Standard Bar After Wearing the Dynamic Bar
Description: On the last day of the study period, parents in the experimental arm were asked in a questionnaire if their child had a hard time returning to the Standard Bar after wearing the Dynamic Bar for approximately 30 days. This was asked to compare parental perception of child comfort in the Dynamic Bar to the Standard Bar.
Time Frame: Study period lasted approximately 90 days.
Population: 7 participants were randomized to the experimental arm to try out the Dynamic Bar.
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Arm
Number analyzed (Participants) | 7
Participants
  Strongly Disagree | 2
  Disagree | 2
  Unsure | 1
  Agree | 2
  Strongly Agree | 0

7. Secondary Outcome: Parental Perception of Child Comfort - Comparison of 5-point Likert Scale Responses
Description: On the first day of the study period, parents in the experimental arm were asked about their child's comfort in the Standard Bar, their child's ability to move their feet/legs normally in the Standard Bar, and their satisfaction with the weight, shape, and size of the Standard Bar.
  Following the study's intervention period, parents in the experimental arm were asked the same questions about the Dynamic Bar.
  Average survey responses were then compared in order to compare parental perception of child comfort in the Dynamic Bar to the Standard Bar.
  Possible survey answers ranged from strongly disagree/very unsatisfied (1) to strongly agree/very satisfied (5). A higher score indicates a more positive perception of the bar.
Time Frame: Intervention period lasted approximately 30 days.
Population: 7 participants were randomized to the experimental arm to try out the Dynamic Bar.
Measure: Mean (Full Range); unit: score on a scale
Groups:
- Experimental Arm Using Standard Bar: Patients were asked about their perception of the Standard Bar at the beginning of the study.
- Experimental Arm Using Dynamic Bar: Patients were asked about their perception of the Dynamic Bar at the end of the study's intervention period.
Arm/Group | Experimental Arm Using Standard Bar | Experimental Arm Using Dynamic Bar
Number analyzed (Participants) | 7 | 7
score on a scale
  Child comfort in bar | 4.3 [3 to 5] | 4.6 [4 to 5]
  Ability to move feet/legs normally in bar | 3.4 [1 to 5] | 4.4 [3 to 5]
  Parent satisfaction with weight of bar | 4.0 [3 to 5] | 3.9 [2 to 5]
  Parent satisfaction with shape of bar | 3.9 [3 to 5] | 4.3 [3 to 5]
  Parent satisfaction with size of bar | 3.9 [2 to 5] | 4.6 [4 to 5]

8. Secondary Outcome: Patient Tolerance of Bracing - Experimental Arm vs. Control Arm - Overall Average
Description: Each patient's brace wear was recorded by parent-report brace logs and iButton temperature sensors in order to compare patient tolerance of the Standard Bar to the Dynamic Bar. For each patient, a bracing adherence fraction was calculated by dividing their average number of daily bracing hours by their prescribed number of daily bracing hours.
  The average adherence fraction in the experimental arm was compared to the average adherence fraction in the control arm during the study's intervention period. Under normal circumstances, the intervention period was the time between the patient's Day 0 visit and Day 30 visit, as that is the period in which patients in the experimental arm should be wearing the Dynamic Bar. However, if a patient in the experimental arm broke the Dynamic Bar and had to return to the Standard Bar during this period, those days were not included in the intervention period.
  This analysis aims to assess if bar type significantly affects bracing tolerance
Time Frame: Intervention period lasted approximately 30 days.
Population: 4 patients completed participation in the control arm, and 7 patients completed participation in the experimental arm. Note that 1 parent in the experimental arm lost their brace wear log during the study's intervention period.
Measure: Mean (Standard Deviation); unit: Average Adherence Fraction
Arm/Group | Control Arm | Experimental Arm
Number analyzed (Participants) | 4 | 7
Average Adherence Fraction
  Parent-reported brace logs: number analyzed (Participants) | 4 | 6
  Parent-reported brace logs | 1.01 (0.14) | 0.97 (0.06)
  iButton temperature sensors | 1.03 (0.15) | 0.91 (0.07)
Statistical Analysis 1: Comparison: Control Arm vs Experimental Arm; The null hypothesis is that there is no difference in brace adherence fractions between the control arm and the experimental arm during the study's intervention period. In this test, brace wear was measured by parent-reported brace logs; Test type: Equivalence — This analysis uses Welch's t-tests to calculate statistical significance, given the different variances and sample sizes of the populations; p = 0.67, t-test, 2 sided — The threshold for statistical significance was p = 0.05; Degrees of Freedom = 3.82
Statistical Analysis 2: Comparison: Control Arm vs Experimental Arm; The null hypothesis is that there is no difference in brace adherence fractions between the control arm and the experimental arm during the study's intervention period. In this test, brace wear was measured by iButton temperature sensors; Test type: Equivalence — [test comment as in outcome 8, analysis 1]; p = 0.23, t-test, 2 sided — The threshold for statistical significance was p = 0.05; Degrees of Freedom = 3.70

9. Secondary Outcome: Patient Tolerance of Bracing - Dynamic Bar vs. Standard Bar (Experimental Arm Only) - Overall Average
Description: Each patient's brace wear was recorded by parent-report brace logs and iButton temperature sensors in order to compare patient tolerance of the Standard Bar to the Dynamic Bar. For each patient, a bracing adherence fraction was calculated by dividing their average number of daily bracing hours by their prescribed number of daily bracing hours.
  Since patients in the experimental arm used both the Dynamic Bar and the Standard Bar during the study period, their average adherence fraction when wearing the Dynamic Bar was compared to their average adherence fraction when wearing the Standard Bar over the entire study period.
  This analysis aims to assess if bar type significantly affects bracing tolerance.
Time Frame: Experimental arm used the Dynamic Bar for approximately 30 days, then used the Standard Bar for approximately 60 days
Population: 7 patients completed participation in the experimental arm. Note that 2 of these parents lost their brace wear logs when their child was wearing the Standard Bar, and 1 of these parents lost their brace wear log when their child was wearing the Dynamic Bar.
Measure: Mean (Standard Deviation); unit: Average Adherence Fraction
Groups:
- Experimental Arm Using the Standard Bar: This group represents the time period in which the experimental arm was wearing the Standard Bar during the study period.
- Experimental Arm Using the Dynamic Bar: This group represents the time period in which the experimental arm was wearing the Dynamic Bar during the study period.
Arm/Group | Experimental Arm Using the Standard Bar | Experimental Arm Using the Dynamic Bar
Number analyzed (Participants) | 7 | 7
Average Adherence Fraction
  Parent-reported brace logs: number analyzed (Participants) | 5 | 6
  Parent-reported brace logs | 0.96 (0.09) | 0.97 (0.06)
  iButton temperature sensors | 0.78 (0.24) | 0.91 (0.07)
Statistical Analysis 1: Comparison: Experimental Arm Using the Standard Bar vs Experimental Arm Using the Dynamic Bar; The null hypothesis is that there is no difference in brace adherence fractions when the experimental arm is wearing the Dynamic Bar versus the Standard Bar during the study period. In this test, brace wear was measured by parent-reported brace logs; Test type: Equivalence — [test comment as in outcome 8, analysis 1]; p = 0.86, t-test, 2 sided — The threshold for statistical significance was p = 0.05; Degrees of Freedom = 6.68
Statistical Analysis 2: Comparison: Experimental Arm Using the Standard Bar vs Experimental Arm Using the Dynamic Bar; The null hypothesis is that there is no difference in brace adherence fractions when the experimental arm is wearing the Dynamic Bar versus the Standard Bar during the study period. In this test, brace wear was measured by iButton temperature sensors; Test type: Equivalence — [test comment as in outcome 8, analysis 1]; p = 0.21, t-test, 2 sided — The threshold for statistical significance was p = 0.05; Degrees of Freedom = 6.94

10. Secondary Outcome: Patient Tolerance of Bracing - Dynamic Bar vs. Standard Bar (Experimental Arm Only) - N of 1
Description: as for outcome 9
Time Frame: Experimental arm used the Dynamic Bar for approximately 30 days, then used the Standard Bar for approximately 60 days
Population: 7 patients completed participation in the experimental arm. Note that 2 of these parents lost their brace wear logs when their child was wearing the Standard Bar, and 1 of these parents lost their brace wear log when their child was wearing the Dynamic Bar. As such, only 5/7 had brace log data in both bar types that could be used in this analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Experimental Arm - Wore the Standard Bar More Than the Dynamic Bar: This group represents the number of patients in the experimental arm who had a higher bracing adherence fraction when wearing the Standard Bar than they did when wearing the Dynamic Bar during the study period.
- Experimental Arm - Wore the Dynamic Bar More Than the Standard Bar: This group represents the number of patients in the experimental arm who had a higher bracing adherence fraction when wearing the Dynamic Bar than they did when wearing the Standard Bar during the study period.
Arm/Group | Experimental Arm - Wore the Standard Bar More Than the Dynamic Bar | Experimental Arm - Wore the Dynamic Bar More Than the Standard Bar
Number analyzed (Participants) | 7 | 7
Participants
  Parent-reported brace logs: number analyzed (Participants) | 5 | 5
  Parent-reported brace logs | 2 | 3
  iButton temperature sensors | 2 | 5

11. Secondary Outcome: Number of Clubfoot Recurrences During the Study Period
Description: All clubfoot recurrences that occurred during the study period were tracked to perform a preliminary assessment of the effectiveness of the Dynamic Bar at preventing clubfoot recurrence.
  For this analysis, clubfoot recurrence was pre-defined as a Pirani score > 0.5, a new occurrence of cavus, adduction and/or hindfoot varus, or a loss of passive ankle dorsiflexion (equinus) of < 10 degrees above neutral or a reduction of 5 or more degrees from the previous visit. All adverse adverse events that were deemed "unrelated" to the foot abduction bar, per the blinded outcomes assessor, were omitted from this analysis.
  The null hypothesis is that 'the Dynamic Bar does not lead to higher rates of clubfoot recurrence,' and it will be rejected if the number of patients who wore their FAB as prescribed and develop clubfoot recurrence, is substantially greater in the experimental arm than it is in the control arm (i.e. a difference of more than 2 cases).
Time Frame: Study period lasted approximately 90 days.
Population: All parents self-reported fair compliance to the prescribed bracing schedule (within 1 hour of the prescribed bracing range per day). However, the sensors reported that 3 patients wore the brace much less than prescribed during the study (deficit of >1.5 hours/day).
  Note that all AEs related to recurrence were classified as non-serious, mild, and not unexpected, and therefore may not represent a true relapse in clubfoot treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Control Arm | Experimental Arm
Number analyzed (Participants) | 4 | 7
Participants
  All patients | 2 | 0
  Patients with fair brace compliance per logs and sensors (+/- 1 hr of the prescribed range per day): number analyzed (Participants) | 3 | 5
  Patients with fair brace compliance per logs and sensors (+/- 1 hr of the prescribed range per day) | 1 | 0

12. Other Pre Specified Outcome: Video Data Analysis - Comparing the Range of Motion Provided by the Dynamic Bar vs. Standard Bar
Description: Parents were given the option of consenting to video recordings being taken of the patient's feet and legs while wearing their prescribed bar. These videos were closely studied to compare the range of motion provided by the Standard Bar to the Dynamic Bar, and to verify that the Dynamic Bar consistently maintains proper foot position and leg alignment during use.
Time Frame: Each video recording was approximately 2 minutes in length.
Population: All participants consented to video recording.
Measure: Count of Participants; unit: Participants
Groups:
- Control Arm Using Standard Bar: This group continued using the Standard Bar as part of their brace, per their current treatment.
- Experimental Arm Using Dynamic Bar: This group used the Dynamic Bar for 30 days instead of their Standard Bar.
Arm/Group | Control Arm Using Standard Bar | Experimental Arm Using Dynamic Bar
Number analyzed (Participants) | 4 | 7
Participants
  Patients that were noted to achieve normal developmental motor skills during video recording. | 4 | 7
  Patients that were noted to achieve intermittent ankle plantarflexion during video recording. | 1 | 2

13. Post Hoc Outcome: Breakages and Malfunctions of the Dynamic Bar Prototype
Description: To refine the design of the Dynamic Bar prototype for future use, the study team documented all bar breakages/malfunctions that occurred during the study period.
Time Frame: Each patient in the experimental arm used the Dynamic Bar for approximately 30 days. Most Dynamic Bars were only used by one patient, but two Dynamic Bars were used by two patients each.
Population: The first two breakages/malfunctions identified below resulted in the immediate suspension of the Dynamic Bar prototypes until the bars could be redesigned.
  The last three breakages/malfunctions identified below are specific to the latest version of the Dynamic Bar, which was used on all 7 participants in the experimental arm.
Measure: Number; unit: cases observed
Groups:
- Breakages and Malfunctions of the Dynamic Bar: Breakages and malfunctions that occurred to the Dynamic Bar prototypes during the study period.
Arm/Group | Breakages and Malfunctions of the Dynamic Bar
Number analyzed (Participants) | 7
cases observed
  Participant pinched their finger in the pin-slot mechanism (this prompted immediate bar redesign) | 1
  Ball joint popped out of socket in ball joint linkage (this prompted immediate bar redesign) | 3
  End caps on the L brackets were torn by the participant | 2
  Crossbar snapped in two | 1
  Wear was observed on the brass components in the ball joint linkages | 6

ADVERSE EVENTS:
Time Frame: Adverse Event (AE) data was collected at each study visit over the entire study period, which lasted for approximately 3 months per participant.
Description: AEs were classified as: Serious or non-serious; Mild, moderate, or severe; Unexpected or not unexpected; Unrelated, unlikely to be related, possibly related, probably related, or definitely related to the bar.
  It is not appropriate to separate the 'Experimental Arm wearing the Dynamic Bar' from the 'Experimental Arm wearing the Standing Bar' because the study period is short and there is potential for late-onset AEs. (AEs may have been caused by the Dynamic Bar but were only noted on Day 90.)
Groups:
- Experimental Arm Using Experimental Bar Then Standard Bar: This group used the Dynamic Bar for 30 days then returned to their Standard Bar for 60 days.
Arm/Group | Control Arm Using Standard Bar | Experimental Arm Using Experimental Bar Then Standard Bar
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/7
Other Adverse Events (participants affected / at risk) | 3/4 | 4/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Arm Using Standard Bar (N=4) | Experimental Arm Using Experimental Bar Then Standard Bar (N=7)
Pressure sore, skin rash, and/or redness (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (4) — Classified as mild and not unexpected. 2/4 cases that occurred in the experimental arm were deemed unrelated to the Dynamic Bar arm per the blinded outcomes assessor (likely related to new clubfoot boots).
Pinched finger in foot abduction bar (Product Issues) | 0 (0) | 1 (1) — Classified as mild and unexpected. Parent reported that patient pinched their finger inside a slot in the Dynamic Bar, resulting in minor redness. This prompted immediate suspension of the Dynamic Bar for all participants until the slot was removed.
Development of mild MTP adduction (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) — Classified as mild and not unexpected. The case of MTP adduction that occurred in the experimental arm was deemed unrelated to the use of the Dynamic Bar per the blinded outcomes assessor (adduction previously noted in patient's chart).
Development of mild dynamic supination (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Classified as mild and not unexpected.
Decreased eversion strength (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Classified as mild and not unexpected.
Decreased passive dorsiflexion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Classified as mild and not unexpected. Consisted of a 5 degree decrease in passive dorsiflexion during the study period, but remains well within normal range.
Decreased external foot progression angle (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Classified as mild and not unexpected. Consisted of a 5-10 degree decrease in external foot progression angle during the study period.

LIMITATIONS AND CAVEATS:
Recruitment closed early, due to limited hospital resources, leading to a small number of subjects analyzed.

Several large discrepancies were noted between the iButton sensor data and the brace log data. This calls into question the reliability of iButton sensors in accurately measuring brace wear in clubfoot treatment. Additionally, the sensors only recorded the temperature every 45 minutes due to limited data storage; this increases the error associated with the brace wear calculations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-04): https://cdn.clinicaltrials.gov/large-docs/43/NCT05293743/Prot_SAP_000.pdf